CLINICAL TRIAL: NCT03079726
Title: Use of Device Data to Predict Frailty in Individuals With Cardiovascular Implantable Electrical Devices: Pilot Study
Brief Title: Use of Device Data to Predict Frailty in Individuals
Acronym: FRAILCIED
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 16-2587
Record Dates: First submitted 2017-03-06; First posted 2017-03-14 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Age Problem; Morality; Arrhythmias, Cardiac
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Frail individuals (case): Individuals classified as frail based on several clinical metrics
- Non-frail individuals: Individuals failing to meet criteria for frailty based on clinical metrics

SUMMARY:
This is an investigation to examine the correlation and predictive ability of activity measures obtained from cardiovascular implantable electrical devices.

DETAILED DESCRIPTION:
Technology is providing new opportunities to gain insight into patient health in a manner far superior to what can be obtained from routine office visits. For geriatric patients, frailty is one such measure, which has been shown to have a negative correlation with outcomes, including hospitalizations, complications following invasive procedures, and overall mortality. Methods to quantify frailty have been highly limited and somewhat controversial, largely because of their cross-sectional nature. Efforts to obtain longitudinal measures of frailty using activity monitors and other wearable devices have been promising, although they are limited by patient cooperation and cost.

In addition to their therapeutic functions, cardiovascular implantable electrical devices (CIEDs) collect large amounts of data on individuals in whom they are implanted, which can be accessed during office visits as well as remotely. Importantly, the data is obtained passively and routinely from all patients, requiring little to no additional effort or expense. The possibility that activity measures from CIEDs could be used to evaluate frailty, as well as other outcomes, would provide a powerful tool for clinicians to apply data science directly to patients.

This pilot investigation will assess the feasibility of using CIED-derived activity data to predict frailty, and other outcomes, in older populations. The investigators plan to enroll subjects in whom CIEDs are implanted from the University of Colorado Hospital Device clinic, and analyze their data to assess the correlation of daily activity with frailty measures, as well as with cardiac and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Individuals followed in the UCH device clinic
* Individuals with CIED implanted
* Age over 65

Exclusion Criteria:

* Unable/unwilling to provide informed consent

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The investigators plan to enroll all individuals followed in the UCH device clinic, in whom CIED data is available for analysis who are over age 65, and willing and able to provide informed consent. We will not a priori exclude individuals unable to take part in the walk-time, survey/questionnaire assessment, or mini-Cog assessment, although these individuals may be excluded during analysis.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-09-07 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Changes in Daily Activity as measured with a Cardiovascular Implantable Electrical Device (CIED) | 30 - 180 days
  Daily activity adjudicated by CIED algorithm
Presence of Cardiac arrhythmias | From study onset until 2 years
  Any atrial or ventricular arrhythmia
Hospitalizations and Mortality | From study onset until 2 years
  Any hospitalization or death

CONTACTS AND LOCATIONS:
Overall Officials: Michael Rosenberg, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Denver, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided
Plan for initial analysis; sharing if appropriate de-identification is determined possible by IRB and co-investigators